CLINICAL TRIAL: NCT05550844
Title: Frequency and Characteristics of Emphysema in Patients With a FLNA Gene Mutation
Brief Title: EMPHYSEMA AND FLNA MUTATION
Acronym: E-FNLA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Santelys Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0511; 2022-A00972-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2022-09

CONDITIONS: Emphysema
Keywords: Emphysema; Lung function; Filamin A
MeSH Terms: conditions — Emphysema | interventions — Hematologic Tests; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood if emphysema is identified to look for known causes of emphysema (Alpha-1 antitrypsin deficiency, PTPN6 mutation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Chest HRCT — A chest HRCT to identify emphysema
Genetic: blood analysis — If emphysema is identified, a blood analysis will be performed to exclude known causes of emphysema (Alpha-1 antitrypsin deficiency, PTPN6 mutation)
Other: Lung function tests — Lung function tests will be performed in accordance with ATS/ERS technical standard

SUMMARY:
Some sparse scientific data support the hypothesis that otherwise unexplained emphysema may be associated with FLNA mutation. This prospective, monocentric, cross-sectional study aimed to describe the frequency of emphysema in patients carrying an FLNA mutation. Patients with FLNA mutations who accept the study will benefit from a chest physician's clinical examination, respiratory function tests and a chest scan. The primary endpoint is to describe emphysema's frequency in patients carrying FLNA mutation. The other objectives are to describe emphysema's features in these patients and to describe their lung function abnormalities. The final goal is to confirm the association between unexplained emphysema and FLNA mutation.

ELIGIBILITY:
Inclusion Criteria:

* patients with an FLNA mutation (or gene alteration)
* patient who has given written consent to participate in the trial
* socially insured patient
* patient willing to comply with all study procedures and duration

Exclusion Criteria:

* Patient refused or unable to give informed consent
* Administrative reasons: inability to receive information, inability to participate in the entire study, lack of coverage by the social security system,
* Pregnant or breastfeeding women
* Patient under guardianship
* Persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients carrying FLNA mutation identified in Lille University Hospital in BAMARA registry
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Frequency of emphysema in patients carrying FLNA mutation | Baseline
  The presence or absence of emphysema is determined by the chest CT scan.

SECONDARY OUTCOMES:
Morphological of emphysema | Baseline
  type of emphysema: centrilobular/panlobular/mixed
Topographical characteristics of emphysema | Baseline
  predominant distribution of emphysema: upper regions/lower regions/no predominance
The severity of emphysema | Baseline
  objective quantification of emphysema: % of lung volume occupied by emphysema (% of lung with density<-950 HU, 15th percentile parenchyamal density); use of quantification software, available in clinical routine (eXamine; Siemens Healthineers)
Descriptive analysis of functional respiratory abnormalities measured by the functional respiratory test | Baseline
Frequency of unexplained emphysema in patients carrying a FLNA mutation | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Lille University Hospital, Lille, Hauts-de-France, France

REFERENCES:
- [Derived] Michalski A, Vincent-Delorme C, Demoulin-Alexikova S, Smol T, Felloni P, Le Rouzic O, Perez T, Bautin N, Wemeau L, Balduyck M, Zerimech F, Pontana F, Delsart P, Cailliau E, Chenivesse C, Valentin V. Frequency and characteristics of emphysema in adults with FLNA variants: a single-center study. Orphanet J Rare Dis. 2025 Nov 5;20(1):560. doi: 10.1186/s13023-025-04068-6. PMID 41194194